CLINICAL TRIAL: NCT05213884
Title: A Phase II Trial of Induction and Adjuvant Camrelizumab Combined With Chemoradiation in Patients With Locally Advanced Head and Neck Squamous Cell Carcinoma
Brief Title: The Efficacy of Induction and Adjuvant Camrelizumab Combined With Chemoradiation for LA-HNSCC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chongqing University Cancer Hospital (Other)
Responsible Party: Principal Investigator, Ying Wang, Associate Director of Chongqing University Cancer Hospital, Chongqing University Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRIA
Record Dates: First submitted 2022-01-16; First posted 2022-01-28 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Head and Neck Squamous Cell Carcinoma
Keywords: Camrelizumab; Locally Advanced HNSCC; Chemoradiotherapy
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — camrelizumab; spartalizumab; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Camrelizumab plus chemoradiotherapy (Experimental): Induction camrelizumab therapy at least one cycle (every 3 weeks) followed by definitive concurrent chemoradiotherapy. After 4~6 weeks of the completion of radiotherapy, adjuvant camrelizumab therapy will begin every 3 weeks for 16 cycles (1 year) or continue until progression or unacceptable toxicity.
  Interventions: Drug: Camrelizumab; Drug: Concurrent cisplatin chemotherapy; Radiation: Intensity-modulated radiotherapy (IMRT)

INTERVENTIONS:
Drug: Camrelizumab — 200 mg, intravenous infusion over 30 minutes (Q3W); 1~3 cycles of camrelizumab before radiotherapy and camrelizumab are maintained for 16 cycles (1 year) after the end of radiotherapy.
  Other Names: Anti-PD-1 antibody
Drug: Concurrent cisplatin chemotherapy — cisplatin is given at a dose of 40 mg/m2 via intravenous infusion during radiotherapy and starts on the 1st day of radiotherapy every week for 6 cycles.
Radiation: Intensity-modulated radiotherapy (IMRT) — 70 Gy/ 35 fractions/7 weeks, 5 fractions/week, 1 fraction/day.

SUMMARY:
This is a phase 2, single-arm clinical trial, with the purpose to evaluate the therapeutic efficacy and safety of PD-1 Blockade camrelizumab combined with induction chemotherapy followed by concurrent chemoradiotherapy and as adjuvant monotherapy in patients with locally advanced head and neck squamous cell carcinoma.

DETAILED DESCRIPTION:
All participants from 3 hospitals will receive induction camrelizumab therapy at least one cycle (every 3 weeks) followed by definitive concurrent chemoradiotherapy. After 4~6 weeks of the completion of radiotherapy, adjuvant camrelizumab therapy will begin every 3 weeks for 16 cycles (1 year) or continue until progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females ≥18 years of age.
2. ECOG Performance Status 0 or 1.
3. Histological diagnosis of squamous cell carcinoma of the lip, oral cavity, oropharynx, hypopharynx, larynx or nasal sinus.
4. Stage III, IVa, IVb (according to the 8th AJCC edition); Stage III for HPV positive oropharyngeal disease.
5. Inoperable or refused surgery; eligible for definitive concurrent chemoradiotherapy.
6. With measurable target lesions by CT or MRI.
7. Adequate bone marrow function.
8. Adequate renal and liver function.
9. Pregnancy test (for patients of childbearing potential) negative at screening.
10. Signed Written Informed Consent.

Exclusion Criteria:

1. Have a history of immunodeficiency, or have other acquired or congenital immunodeficiency diseases, or have a history of organ transplantation.
2. Active autoimmune disease (Such as type I diabetes, vitiligo, psoriasis, patients who do not need immunosuppressive drugs do not need to be excluded).
3. Has abnormal thyroid function, and the thyroid function cannot be maintained normal despite medical treatment.
4. Pregnancy or breast feeding.
5. Has a history of psychiatric substance abuse, alcoholism, or drug addiction.
6. Prior therapy with a PD-1, anti-PD-Ligand 1 (PD-L1) or CTLA-4 agent.
7. Has received a live vaccine within 4 weeks of planned start of study therapy.
8. Has hepatitis B surface antigen (HBsAg) positive with HBV DNA copy number of ≥1000cps/ml or hepatitis C virus (HCV) antibody positive.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
EFFICACY Progress-free survival (PFS) | 2 years
  Defined as time from randomization to locoregional or distant metastasis relapse or death from any cause, whichever occurred first.

SECONDARY OUTCOMES:
EFFICACY Overall survival (OS) | 2 years
  Overall survival is measured from day of diagnosis until death due to any cause or the latest known date alive.
EFFICACY Objective response rate (ORR） | 2 years
  Defined as a complete response (CR) or partial response (PR) from enrolled until disease progression or death due to any cause.
EFFICACY Duration of response (DOR) | 2 years
  Defined as the time from the first assessment of CR or PR to the first assessment of disease progression or death due to any cause.
SAFETY Incidence rate of adverse events (AEs) | 2 years
  Analysis of adverse events (AEs) are based on treatment-related AEs (trAEs) and immune-related AEs (irAEs), and all-grade AEs and grade 3-4 AEs, according to the Common Terminology Criteria for Adverse Events, version 5.0.
QUALITY OF LIFE Quality of life (QoL): questionnaire | 2 years
  QoL is evaluated with the use of the head-and-neck-specific module (H&N35) of the Quality of Life Questionnaire-Core 30 module (QLQ-C30).

CONTACTS AND LOCATIONS:
Overall Officials: Ying Wang, Ph.D, M.D., Principal Investigator — Chongqing University Cancer Hospital
Locations (3):
- China (3):
  - Chongqing University Cancer Hospital, Chongqing, Chongqing Municipality
  - Chongqing University Three Gorges Hospital, Wanzhou, Chongqing Municipality
  - The Affiliated Hospital of Southwest Medical University, Luzhou, Sichuan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ang KK, Zhang Q, Rosenthal DI, Nguyen-Tan PF, Sherman EJ, Weber RS, Galvin JM, Bonner JA, Harris J, El-Naggar AK, Gillison ML, Jordan RC, Konski AA, Thorstad WL, Trotti A, Beitler JJ, Garden AS, Spanos WJ, Yom SS, Axelrod RS. Randomized phase III trial of concurrent accelerated radiation plus cisplatin with or without cetuximab for stage III to IV head and neck carcinoma: RTOG 0522. J Clin Oncol. 2014 Sep 20;32(27):2940-50. doi: 10.1200/JCO.2013.53.5633. PMID 25154822
- [Background] Seiwert TY, Burtness B, Mehra R, Weiss J, Berger R, Eder JP, Heath K, McClanahan T, Lunceford J, Gause C, Cheng JD, Chow LQ. Safety and clinical activity of pembrolizumab for treatment of recurrent or metastatic squamous cell carcinoma of the head and neck (KEYNOTE-012): an open-label, multicentre, phase 1b trial. Lancet Oncol. 2016 Jul;17(7):956-965. doi: 10.1016/S1470-2045(16)30066-3. Epub 2016 May 27. PMID 27247226
- [Background] Bauml J, Seiwert TY, Pfister DG, Worden F, Liu SV, Gilbert J, Saba NF, Weiss J, Wirth L, Sukari A, Kang H, Gibson MK, Massarelli E, Powell S, Meister A, Shu X, Cheng JD, Haddad R. Pembrolizumab for Platinum- and Cetuximab-Refractory Head and Neck Cancer: Results From a Single-Arm, Phase II Study. J Clin Oncol. 2017 May 10;35(14):1542-1549. doi: 10.1200/JCO.2016.70.1524. Epub 2017 Mar 22. PMID 28328302
- [Background] Lee NY, Ferris RL, Psyrri A, Haddad RI, Tahara M, Bourhis J, Harrington K, Chang PM, Lin JC, Razaq MA, Teixeira MM, Lovey J, Chamois J, Rueda A, Hu C, Dunn LA, Dvorkin MV, De Beukelaer S, Pavlov D, Thurm H, Cohen E. Avelumab plus standard-of-care chemoradiotherapy versus chemoradiotherapy alone in patients with locally advanced squamous cell carcinoma of the head and neck: a randomised, double-blind, placebo-controlled, multicentre, phase 3 trial. Lancet Oncol. 2021 Apr;22(4):450-462. doi: 10.1016/S1470-2045(20)30737-3. PMID 33794205
- [Background] Uppaluri R, Campbell KM, Egloff AM, Zolkind P, Skidmore ZL, Nussenbaum B, Paniello RC, Rich JT, Jackson R, Pipkorn P, Michel LS, Ley J, Oppelt P, Dunn GP, Barnell EK, Spies NC, Lin T, Li T, Mulder DT, Hanna Y, Cirlan I, Pugh TJ, Mudianto T, Riley R, Zhou L, Jo VY, Stachler MD, Hanna GJ, Kass J, Haddad R, Schoenfeld JD, Gjini E, Lako A, Thorstad W, Gay HA, Daly M, Rodig SJ, Hagemann IS, Kallogjeri D, Piccirillo JF, Chernock RD, Griffith M, Griffith OL, Adkins DR. Neoadjuvant and Adjuvant Pembrolizumab in Resectable Locally Advanced, Human Papillomavirus-Unrelated Head and Neck Cancer: A Multicenter, Phase II Trial. Clin Cancer Res. 2020 Oct 1;26(19):5140-5152. doi: 10.1158/1078-0432.CCR-20-1695. Epub 2020 Jul 14. PMID 32665297
- [Background] Zandberg DP, Strome SE. The role of the PD-L1:PD-1 pathway in squamous cell carcinoma of the head and neck. Oral Oncol. 2014 Jul;50(7):627-32. doi: 10.1016/j.oraloncology.2014.04.003. Epub 2014 May 10. PMID 24819861
- [Background] Yang Y, Qu S, Li J, Hu C, Xu M, Li W, Zhou T, Shen L, Wu H, Lang J, Hu G, Luo Z, Fu Z, Qu S, Feng W, Chen X, Lin S, Zhang W, Li X, Sun Y, Lin Z, Lin Q, Lei F, Long J, Hong J, Huang X, Zeng L, Wang P, He X, Zhang B, Yang Q, Zhang X, Zou J, Fang W, Zhang L. Camrelizumab versus placebo in combination with gemcitabine and cisplatin as first-line treatment for recurrent or metastatic nasopharyngeal carcinoma (CAPTAIN-1st): a multicentre, randomised, double-blind, phase 3 trial. Lancet Oncol. 2021 Aug;22(8):1162-1174. doi: 10.1016/S1470-2045(21)00302-8. Epub 2021 Jun 23. PMID 34174189
- [Background] Burtness B, Harrington KJ, Greil R, Soulieres D, Tahara M, de Castro G Jr, Psyrri A, Baste N, Neupane P, Bratland A, Fuereder T, Hughes BGM, Mesia R, Ngamphaiboon N, Rordorf T, Wan Ishak WZ, Hong RL, Gonzalez Mendoza R, Roy A, Zhang Y, Gumuscu B, Cheng JD, Jin F, Rischin D; KEYNOTE-048 Investigators. Pembrolizumab alone or with chemotherapy versus cetuximab with chemotherapy for recurrent or metastatic squamous cell carcinoma of the head and neck (KEYNOTE-048): a randomised, open-label, phase 3 study. Lancet. 2019 Nov 23;394(10212):1915-1928. doi: 10.1016/S0140-6736(19)32591-7. Epub 2019 Nov 1. PMID 31679945